CLINICAL TRIAL: NCT03110640
Title: A Phase I Study of Administrating CD19 Chimeric Antigen Receptor Expressing T Cells Followed by Allogeneic Stem Cell Transplantation in Patients With Refractory CD19+ B-linage Leukemia/Lymphoma
Brief Title: Anti-CD19 CAR T Infusion Combined With Allogeneic Stem Cell Transplantation for B-cell Leukemia/Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Hrain Biotechnology Co., Ltd. (Industry); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Kang YU, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170316
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Hematopoietic/Lymphoid Cancer; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD9CAR-T transfer (Experimental): All subjects will receive allogeneic stem cell transplantation after infusion of αCD19-TCRz-CD28 CAR-T
  Interventions: Biological: anti-CD19 CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19 CAR-T — Ex vivo-expanded autologous T cells modified to express CD19 CAR
Drug: Fludarabine — Patients were given cyclophosphamide 500mg/m2/day on day -4 and fludarabine at 25 mg/m2/day on day -4, day -3, and day -2.
Drug: Cyclophosphamide — Patients were given cyclophosphamide 500mg/m2/day on day -4.

SUMMARY:
This is a single-arm open-label phase I study to determine the effect of CD19- CAR-T Cells infusion followed by allogeneic stem cell transplantation in safety, efficacy and engraftment potential in patients with CD19+ B-lineage leukemia and lymphoma.

DETAILED DESCRIPTION:
Primary objectives

1. To determine the safety and feasibility of allogeneic stem cell transplantation combined with adoptive transfer of T cells modified to express CD19-specific chimeric antigen receptor (CD19CAR) for treatment of leukemia and lymphoma Secondary objectives
2. To measure the efficacy of the CD19CAR T cell infusion combined with allogeneic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

* 5 Years to 70 Years, Male and female;
* Expected survival > 12 weeks;
* Performance score 0-2;
* Histologically confirmed as CD19-positive lymphoma/leukemia and who meet one of the following conditions; Patient receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment; Disease recurrence after stem cell transplantation; Diagnosis as lymphoma, but refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy
* Creatinine < 2.5 mg/dl;
* ALT/AST < 3x normal;
* Bilirubin < 2.0 mg/dl;
* Adequate venous access for apheresis, and no other contraindications for leukapheresis;
* Take contraceptive measures before recruit to this trial;
* Written voluntary informed consent is given.

Exclusion Criteria:

* Patients with symptoms of central nervous system
* Accompanied by other malignant tumor
* Active hepatitis B or C, HIV infection
* Any other diseases could affect the outcome of this trial
* Suffering severe cardiovascular or respiratory disease
* Poorly controlled hypertension
* A history of mental illness and poorly controlled
* Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration
* Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
* Reaching a steady dose if receiving anticoagulant therapy before assignment
* Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Pregnant or lactating women
* Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Safety - incidence of adverse events defined as dose-limited toxicity | 180 days
  incidence of adverse events defined as dose-limited toxicity

SECONDARY OUTCOMES:
Overall complete remission rate | 1 year
  Overall complete remission rate
Duration of remission | 1 year
  Duration of remission

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, M.D., Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affilicated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dong R, Jiang S, Chen Y, Ma Y, Sun L, Xing C, Zhang S, Yu K. Prognostic Significance of Cytokine Release Syndrome in B Cell Hematological Malignancies Patients After Chimeric Antigen Receptor T Cell Therapy. J Interferon Cytokine Res. 2021 Dec;41(12):469-476. doi: 10.1089/jir.2021.0057. PMID 34935483